CLINICAL TRIAL: NCT07165392
Title: Analysis of Neuromodulation as a Complementary Treatment to Evidence-based Clinical Intervention in Subjects With Musculoskeletal Pathology of the Upper Limb: a Double-blind Randomized Clinical Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Dr. Manuel González-Sánchez, Principal Investigator, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 152/2025
Record Dates: First submitted 2025-09-02; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Neuromodulation; Upper Limb; Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases | interventions — Transcutaneous Electric Nerve Stimulation; Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Neuromodulation 2 times per week (Experimental)
  Interventions: Other: Neuromodulation; Other: Physical Exercise; Other: Stretching
- Neuromodulation 3 times per week (Experimental)
  Interventions: Other: Neuromodulation; Other: Physical Exercise; Other: Stretching
- Non-neuromodulation 2 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching
- Non-neuromodulation 3 times per week (Experimental)
  Interventions: Other: Physical Exercise; Other: Stretching

INTERVENTIONS:
Other: Neuromodulation — The application of neuromodulation therapy will be carried out with the support of ultrasound visualization on the anatomical area of the target nerve, seeking a motor and/or sensory response with its stimulation.
  Arms: Neuromodulation 2 times per week; Neuromodulation 3 times per week
Other: Physical Exercise — The therapeutic physical exercise will consist of 3 periods of isometric contraction of 30 seconds, with a rest period of 1 minute, varying the number of repetitions from 3 to 5 depending on the patient's symptoms.
Other: Stretching — To stretch the muscles involved, 3 periods of maximum tolerable stretching without pain will be performed, lasting 20 seconds and resting for 30 seconds.

SUMMARY:
This project aims to analyze the use of neuromodulation within a treatment protocol for musculoskeletal conditions of the upper limb, as well as to determine the difference between two and three sessions per week. Study participants will be divided into four intervention groups: the first will receive two sessions per week for a period of six months, while the second will receive three sessions per week for the same period. The treatment protocol will consist of therapeutic physical exercise focused on the muscles and joints of the lower limb, stretching of the involved muscles, and neuromodulation of the brachial plexus nerve root, which innervates the affected structures. The third and fourth intervention groups will receive the same treatment as mentioned above, but without neuromodulation. The third group will receive three sessions per week, while the second group will receive two sessions per week. Two different types of measurement variables will be used: objective variables will be used to measure range of motion and muscle strength. Subjective variables will also be used through validated questionnaires, covering physical activity, health-related quality of life, upper limb function, and a visual analog scale for pain perception.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the study will be men and women of working age, diagnosed with musculoskeletal disorders of the upper limb, and who have not yet received physical therapy.

Exclusion Criteria:

* Have undergone surgery.
* Those who refuse to participate in this study.
* Patients who present muscular atrophy in the upper limb due to a pathology of the latter.
* Medical conditions that are contraindications for neuromodulation therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
EUROQOL-5D (EQ-5D) | Baseline and up to one year
  It consists of a generic instrument for measuring health-related quality of life (HRQoL), which consists of two parts: a descriptive system for assessing health status (ranging from 1, meaning "I have no problems" to 3, "many problems") and a visual analogue scale (ranging from 0, which is the worst imaginable health status, to 100, which is the best imaginable health status).
SHORT FORM 12 HEALTH SURVEY (SF-12) | Baseline and up to one year
  The SF-12 questionnaire is composed of a subset of 12 items derived from the SF-36, with the physical and mental components being scored as the only items. Depending on the item, response options range from 3 to 6, with each question receiving a value that is subsequently transformed into a scale of 0 to 100. All scores have a mean of 50, with values above or below 50 indicating better or worse health status, respectively, compared to the reference population.
DISABILITIES OF ARM, SHOULDER AND HAND (DASH) | Baseline and up to one year
  It consists of a self-administered questionnaire that assesses the upper limb as a functional unit and allows for the quantification and comparison of the impact of the different processes affecting different regions of the limb. It consists of a core of 30 items and two optional modules with four items each. Each item is scored from 1 to 5, with higher scores corresponding to greater symptom intensity. The final score can range from 30 to 150 points, with a scale of 0 (best possible score) to 100 (worst possible score). The optional modules are scored separately.
UPPER LIMB FUNCTIONAL INDEX (ULFI) | Baseline and up to one year
  This is a 25-item questionnaire that measures upper limb function. Patients are asked to answer YES if they can perform the action (1 point) and NO if they cannot perform it (0 points). There is also a HALF option (partially perform it), which is worth 0.5 points. The score is then obtained by summing the responses and is finally converted into a 100-point percentage scale.
International Physical Activity Questionnaire (IPAQ) | Baseline and up to one year
  An instrument designed to measure physical activity levels in an adult population and serve as a reference for making recommendations regarding physical activity. It comes in two versions: the long version with 31 items (IPAQ-LF) and the short version with 9 items (IPAQ-SF). The short version, which will be used in this study as recommended by the authors, measures activity at four intensity levels, ranging from 1 (vigorous activity) to 4 (sedentary).
Visual Analogue Scale (VAS) | Baseline and up to one year
  It consists of an 11-point numerical scale, ranging from 0 (no pain) to 10 (maximum pain intensity), which serves as a quantification for measuring pain intensity. It has moderate to good reliability.
RANGE OF MOTION | Baseline and up to one year
  Range of motion refers to the number of degrees through which a joint is capable of moving. To measure the elbow's flexion-extension range, the flexion and extension movements are recorded with the arms at the sides and the elbows fully extended. For the forearm, supination and pronation movements are measured with the arm relaxed. For the shoulder, the degrees of flexion, extension, abduction, adduction, and internal and external rotation are measured with the patient in a seated position. Finally, to measure flexion, extension, and radial and ulnar deviations at the wrist, the hand is placed on a flat surface. Measurements are taken with an electronic goniometer, and the patient will be asked to cooperate in determining the pain limit.
MUSCULAR STRENGTH | Baseline and up to one year
  Isometric muscle strength will be assessed using a dynamometer.